CLINICAL TRIAL: NCT06028165
Title: A Prospective, Randomized Comparison of Coronary Artery Bypass Grafting Based on COmputed Tomography-derived Fractional Flow REserve Versus Angiography (CABG-COREA Trial)
Brief Title: CABG Based on CT-FFR Versus Conventional Coronary Angiography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myongji Hospital (Other)
Responsible Party: Principal Investigator, Min-Seok Kim, Associate Professor, Myongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MyongjiH
Record Dates: First submitted 2023-08-29; First posted 2023-09-08 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAG group (Active Comparator): Patients who underwent coronary artery bypass grafting based on conventional coronary angiography (quantitative coronary angiography)
  Interventions: Procedure: Coronary artery bypass grafting based on conventional coronary angiography
- CT-FFR group (Active Comparator): Patients who underwent coronary artery bypass grafting based on cardiac computed tomography-derived fractional flow reserve
  Interventions: Procedure: Coronary artery bypass grafting based on cardiac computed tomography-derived fractional flow reserve.

INTERVENTIONS:
Procedure: Coronary artery bypass grafting based on conventional coronary angiography — Revascularized coronary arteries are decided based on conventional coronary angiography (quantitative coronary angiography)
  Arms: CAG group
Procedure: Coronary artery bypass grafting based on cardiac computed tomography-derived fractional flow reserve. — Revascularized coronary arteries are decided based on cardiac computed tomography-derived fractional flow reserve.
  Arms: CT-FFR group

SUMMARY:
The aims of study are (1) to compare early and 1-year graft patency rates in patients who underwent coronary artery bypass grafting (CABG) based on conventional coronary angiography(CAG) versus cardiac computed tomography(CT)-derived fractional flow reserve(FFR), and (2) to demonstrate difference in clinical outcomes between the 2 groups.

DETAILED DESCRIPTION:
The CABG-COREA trial is designed as a randomized, controlled trial to recruit 96 patients who undergo coronary artery bypass grafting. Patients were randomized by use of a randomization table. Coronary arteries are revascularized based on conventional coronary angiography (quantitative coronary angiography) or cardiac computed tomography-derived fractional flow reserve according to the randomization result.

The primary end point is to evaluate early and 1-year postoperative graft patency. The secondary end points are overall survival, freedom from cardiac death and freedom from MACCE(major adverse cardiac or cerebrovascular events).

ELIGIBILITY:
Inclusion Criteria:

* age equal or more than 40
* age equal or less than 80
* patients who undergo coronary artery bypass grafting due to multi-vessel coronary artery disease
* patients who agree to the enrollment

Exclusion Criteria:

* Patients with heart failure (left ventricular ejection fraction < 25%)
* patients who have intractable ventricular arrhythmia
* patients who has been treated for cancer
* patients who has infectious disease
* patients who are planned to undergo combined cardiac surgery
* patients who has medical co-morbidity with expected survival less than 1 year
* patients with a history of previous cardiac surgery
* Patients with chronic renal failure requiring dialysis
* patients who undergo emergency operation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
1-Year graft patency rates | 1 year
  postoperative graft patency measured by 1 year postoperative coronary angiography

SECONDARY OUTCOMES:
Overall survival | 4 years
  Overall survival rate at 4 years
Freedom from Cardiac Death | 4 years
  Freedom from cardiac death at 4 years
Freedom From MACCE(Major Adverse Cardiac and Cerebrovascular Events) | 4 years
  freedom from MACCE(major adverse cardiac and cerebrovascular events)at 4 years
Early Angiographic Patency Rates | 1.5 days
  The patency rate of the grafts evaluated with coronary angiograms early after coronary artery bypass grafting

CONTACTS AND LOCATIONS:
Overall Officials: Min-Seok Kim, MD, PhD, MSc, Study Chair — Cardiovascular Center, Myongji Hospital
Locations (1):
- Myongji Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.